CLINICAL TRIAL: NCT07020949
Title: Multiple Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Efficacy of THDBH120 in Chinese Patients With T2DM: A Randomized, Bouble-Blind, Placebo-Controlled Phase Ib Trial
Brief Title: Multiple Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Efficacy of THDBH120 in Chinese Patients With T2DM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tonghua Dongbao Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: THDBH120L102
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THDBH120 injection (Experimental)
  Interventions: Drug: THDBH120 injection
- Placebo of THDBH120 injection (Placebo Comparator)
  Interventions: Drug: Placebo of THDBH120 injection

INTERVENTIONS:
Drug: THDBH120 injection — Participants received THDBH120 by subcutaneous injection.
  Arms: THDBH120 injection
Drug: Placebo of THDBH120 injection — Participants received placebo by subcutaneous injection.
  Arms: Placebo of THDBH120 injection

SUMMARY:
The aim of this trial is to investigate the safety, tolerability, pharmacokinetics, and efficacy of THDBH120 injection in participants with T2DM. This study includes three multiple-ascending dose cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 to 75 years of age, inclusive;
* Have T2DM for at least 6 months before screening based on the disease diagnostic criteria (World Health Organization [WHO] Classification for Diabetes);
* Treated with diet and exercise alone, or a stable dose of metformin (≥1000 mg/day and not more than the locally approved dose) for at least 2 months prior to screening;
* Have a BMI between 23 and 35 kg/m²(inclusive) at screening;
* HbA1c levels: 7.0% to 10.0% (inclusive) for subjects treated by diet or exercise alone; 7.0% to 9.0% (inclusive) for subjects receiving stable-dose metformin.

Exclusion Criteria:

* Have been diagnosed with proliferative diabetic retinopathy, diabetic maculopathy, or non-proliferative diabetic retinopathy requiring treatment during the study;
* Have a personal or family history of medullary thyroid carcinoma or have multiple endocrine neoplasia type 2;
* Have diagnosed hyperthyroidism or hypothyroidism;
* Have grade 2 hypoglycemia events or grade 3 hypoglycemia events within 6 months prior to screening;
* Have a history of ketoacidosis, lactic acidosis, or hyperosmolar state leading to hospitalization within 6 months prior to screening;
* Presence of uncontrolled hypertension at screening: systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg;
* Prolonged QTcF interval on 12-lead ECG at screening (QTcF≥450 ms for males, >470 ms for females), PR interval >200 ms, or the presence of long QT syndrome, second- or third-degree atrioventricular block, left or right bundle branch block, Wolff-Parkinson-White syndrome, or any other clinically significant arrhythmias (except sinus arrhythmia);
* Weight change ≥ 5% within 3 months prior to screening;
* Have been treated with insulin, excluding insulin therapy for gestational diabetes mellitus, or acute/temporary insulin therapy (≤ 14 days) for conditions such as acute illness, hospitalization, or elective surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Adverse Event(s) and Serious Adverse Event(s) | 78 days

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of THDBH120. | Day 1 Pre-dose through Day 43
Pharmacokinetics (PK): Maximum Drug Concentration (Cmax) of THDBH120 | Day 1 Pre-dose through Day 43
Change From Baseline in HbA1C | 43 days
Number of Participants With Anti-THBHD120 Antibodies | 78 days

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No